CLINICAL TRIAL: NCT02309463
Title: A Prospective Multicenter Study to Assess the Correlation of LONGterm Wrist ACTigraphy Recorded Physical Performance and 6-minute Walk Distance in Patients With Pulmonary Arterial Hypertension Newly Initiating Endothelin Receptor Antagonist Therapy
Brief Title: Correlation of LONGterm Wrist ACTigraphy Recorded Physical Performance & 6-minute Walk Distance in Patients With Pulmonary Arterial Hypertension
Acronym: LONGACT
Status: Withdrawn | Type: Observational
Why Stopped: EC did not accept measurement of patient's activity for the primary end-point with a non-validated activity tracking device
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-055-506
Record Dates: First submitted 2014-10-22; First posted 2014-12-05 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Endothelin receptor antagonist therapy

SUMMARY:
The objective of the study is to monitor physical activity longitudinally with a wrist activity tracker specifically in PAH patients newly initiating ERA therapy and to assess the correlation with the 6MWD at different time points. Further objectives are to assess the correlation of physical activity measured with the tracker and other parameters for clinical evaluation and right ventricular function assessment (i.e. Biomarkers, WHO Functional class, hospitalization due to PAH, Echochardiography and Quality of Life) as well as sleep efficacy in PAH patients newly initiating ERA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with right heart catheter (RHC)-confirmed PAH (WHO PH group I)
* Age ≥18 year
* Not receiving ERA therapy in the 30 days prior to the enrolment visit
* Signed patient informed consent form

Exclusion Criteria:

* Patient with conditions that prevent compliance with the protocol or to adhere to therapy and use of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PAH, and not receiving ERA therapy in the 30 days prior to the enrolment visit, are eligible for inclusion in this study. Patients in need of ERA therapy will receive ERA treatment according to the physician's decision
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2016-01-31 (Estimated); Study Completion 2017-02-28 (Estimated)

PRIMARY OUTCOMES:
Activity score measured with an electronic activity tracker and absolute 6MWD assessed at different time points during ERA treatment | Baseline to Week 54
Change of physical activity measured with an electronic activity tracker and 6MWD in PAH patients newly initiating ERA therapy between visit 0 and end of observation | baseline to week 54

SECONDARY OUTCOMES:
WHO Functional Class | Baseline to Week 54
NT-ProBNP/BNP | Baseline to Week 54
Echocardiography parameters | Baseline to Week 54
  * Tricuspid pressure gradient
  * TAPSE
  * Pulmonary outflow tract acceleration time
  * Right ventricular fractional area change
  * Pericardial effusion
Number of hospitalization due to PAH (min. overnight) | Baseline to Week 54
Quality of Life | Baseline to Week 54
  Minnesota Living with Heart Failure Questionnaire (MLHFQ)